CLINICAL TRIAL: NCT03306654
Title: A Randomized Trial Examining the Impact of Three 8-week Online Well-Being Programs on Employment-Related Absenteeism, Engagement, Burnout, Stress, and Resilience
Brief Title: Efficacy of Three Online Well-Being Programs to Improve Work-Related Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Happify Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2.5
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Well-being

STUDY DESIGN:
Intervention Model Description: Users are randomly assigned between arms after completing baseline assessment and stay in that arm for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unchanged Happify (Active Comparator): Participants use Happify as it is currently available to consumers on the main site, including all engagement elements. Users may access a wide variety of 4-week programs and use them in any way they desire for the entire study period.
  Interventions: Behavioral: Happify
- Active control (Placebo Comparator): Participants complete a Happify program that is designed to engage with specific activities, but that does not aim to promote positive emotion or reduce negative emotion. Participants gain access to 8 weeks worth of content, but may repeat the content as often as they like in the follow-up period.
  Interventions: Behavioral: Happify
- Distraction condition (Sham Comparator): Participants complete a series of quizzes and polls on Happify designed to engage them in thinking about well-being topics, but without giving any specific instructions for how to promote well-being. Participants gain access to 8 weeks worth of content, but may repeat the content as often as they like in the follow-up period.
  Interventions: Behavioral: Happify

INTERVENTIONS:
Behavioral: Happify — An online platform for conveying techniques from positive psychology, cognitive-behavioral therapy, and mindfulness-based stress reduction.

SUMMARY:
Participants will be randomly assigned between three well-being programs, and assessed with questionnaires before and after the 8-week program, as well as 1-month after the end of the program.

DETAILED DESCRIPTION:
Participants will be randomly assigned between three different well-being programs, with each program lasting 8-weeks and taking place on a simplified research version of the Happify platform. Well-being programs include the unchanged Happify platform, a version of the Happify platform that is designed to engage with specific activities but does not aim to promote positive emotion or reduce negative emotion (i.e., Placebo condition), and a version of the Happify platform that encourages thinking about well-being through quizzes and polls without providing any instructions for promotion (i.e., Wait-list Control). Participants will be asked to complete questionnaires before and after the 8-week program, as well as a 1-month follow-up questionnaire after the program is complete, at which point study participation will end.

ELIGIBILITY:
Inclusion Criteria:

* No prior experience on the Happify platform (new user registration)
* Full-time employment

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Absenteeism (Health and Performance Questionnaire, HPQ [World Health Organization (WHO), 2002]) | Change from baseline to 8-week post, 1-month follow-up
  An 8-item subset of the HPQ focusing on job absenteeism and work quality. Participants will be asked to indicate how many times in the past week they missed part of/an entire work day due to problems with their physical or mental health, and to indicate how often in the past 7 days the quality of their work suffered (e.g., how often they found themselves not working as carefully as they should).
Work Engagement (Utrecht Work Engagement Scale [Schaufeli et al., 2002]) | Change from baseline to 8-week post, 1-month follow-up
  A 2-item subset of the UWES focusing on job resilience and perseverance. Participants will be asked to indicate how frequently they feel mentally resilient at their job and how frequently they persevere.
Burnout (Maslach Burnout Inventory [Maslach & Jackson, 1981]) | Change from baseline to 8-week post, 1-month follow-up
  A 5-item subset of the MBI focusing on feeling burned out in work settings. Participants will be asked to indicate the extent to which they agree that they feel burned out (e.g., that they feel burned out from their work or feel frustrated by their job).
Job-Related Stress (Stress-related Presenteeism Scale [Gilbreath & Frew, 2008]) | Change from baseline to 8-week post, 1-month follow-up
  A 6-item measure of job stress-related presenteeism. Participants will be asked to indicate how frequently they suffer from stress-related presenteeism is work (e.g., they are unable to concentrate on their job at work, or stress distracts their attention away from job tasks).
Resilience (composite of Perceived Stress Scale [Cohen et al., 1983], Happify Scale [Carpenter et al., 2016] and Life Orientation Scale, Revised [Scheier & Carver, 1985]). | Change from baseline to 8-week post, 1-month follow-up
  Composite score made of perceived stress, positive emotionality, and optimism. Perceived stress was measured using the Perceived Stress Scale (PSS; Cohen, Kamarck, & Mermelstein, 1983), a 10-item questionnaire that asks users to rate on a scale of 0 (never) to 4 (very often) how frequently they experience various symptoms of feeling stress. Positive emotionality was measured using the emotion subscale of the Happify Scale (HS-E; Carpenter, Crutchley, Zilca, Schwartz, Smith, Cobb, & Parks, 2016), which is a 4-item scale asking participants to rate the extent to which, over the past week, they have experienced positive and negative emotions that are activated or de-activated. Optimism was measured using the Life Orientation Scale, Revised (LOT-R; Scheier & Carver, 1985), a 6-item scale on which participants rate the extent to which they identify with optimistic or pessimistic beliefs.
Absenteeism (Healthy Days measure [Center for Disease Control (CDC), 2000]) | Change from baseline to 8-week post, 1-month follow-up
  A 1-item measure of the extent to which poor physical/mental health prevents one from doing their usual activities, such as self-care, work, or recreation, in the past 30 days [CDC, 2002].

CONTACTS AND LOCATIONS:
Locations (1):
- Happify (an online platform -- study is entirely online), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carpenter J, Crutchley P, Zilca RD, Schwartz HA, Smith LK, Cobb AM, Parks AC. Seeing the "Big" Picture: Big Data Methods for Exploring Relationships Between Usage, Language, and Outcome in Internet Intervention Data. J Med Internet Res. 2016 Aug 31;18(8):e241. doi: 10.2196/jmir.5725. PMID 27580524
- See also: Site where study is taking place — http://www.happify.com